CLINICAL TRIAL: NCT01979822
Title: LPS (Lenus Pro Safety) - Study in Pulmonary Hypertension (PH)
Brief Title: LenusPro Safety (LPS) Study in Patients With PH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Prof. Ralf Ewert, M.D., University Medicine Greifswald
Other Study IDs: LPS-1; LPS-1-2013 (Other: University of Greifswald)
Record Dates: First submitted 2013-09-25; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Hypertension
Keywords: medication pump, complications, safety observation
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PH patients with LenusPro pump: Patient Inclusion Criteria:
  1. Patient aged ≥ 18 years;
  2. diagnosed with Pulmonary Arterial Hypertension (WHO) Category Group 1
  3. Patient is in stable clinical condition and
  4. the previous specific PH medication has been retained unchanged during the past 3 weeks
  Interventions: Other: PH patients with LenusPro pump

INTERVENTIONS:
Other: PH patients with LenusPro pump — Observation/measurement of complications in PH patients with LenusPro pump in the frist six month after implantation of pump

SUMMARY:
The clinical study aims to investigate the numbers of predefined complications in the first six month after implantation of the implantable LENUS Pro® medications pump for intravenous application of treprostinil sodium in patients with PAH.

The manufacturer is Tricumed GmbH, Germany; exclusive marketing rights: OMT GmbH & Co KG 78665 Frittlingen, Germany.

DETAILED DESCRIPTION:
The previously used fully implantable pumps have been improved by development of additional safety options (e.g. acoustic occlusion alarm) for use in patients with PH. In the meantime, the pump (manufacturer: Tricumed GmbH, Germany, exclusively marketing rights: OMT GmbH & Co KG, 78665 Frittlingen, Germany) is offered with an option that meets the requirements for use in treating PH patients. It is based on a constant flow system that consists of gas driven micro-infusion via a chip capillary. The medication is filled into a titanium reservoir via a so-called filling septum (silicon membrane). The membrane is punctured percutaneously with a special needle by specially trained personnel for filling under aseptic conditions. Various safety options ensure a continuous flow rate of the medication and signalize any malfunctions. If catheter occlusion is signalized, the catheter can be rinsed through a second septum in the pump after a percutaneous puncture without emptying the medication reservoir. The pump is available in two sizes (20 ml or 40 ml filling volume). The flow rate set for the 20 ml pump is 1.0 ml/ 24 hours, so that refilling is required every 19 to 20 days. The flow rate set for the 40 ml pump is 2.3 ml/ 24 hours, so that refilling is required every 29 to 30 days. Initial experience with the use of this pump has shown good results for up to 3 years of use (minor complications during implantation, no pump defects in long-term usage, reliable filling under outpatient conditions).

R. Ewert; M. Halank, L. Bruch; H.A. Ghofrani. The implantable pump - a new option for intravenous therapy in patients with severe pulmonary hypertension. Am J Respir Crit Care 2012;186:1196-98 Steringer-Mascherbauer R., Eder V., Ebner Ch. et al. First experience with intravenous treprostinil delivered by an implantable pump (Lenus Pro®) with filling intervals of 28 days in a patient with pulmonary arterial hypertension (PAH) - a case report. ATS Poster Desole S, Velik-Salchner C, Fraedrich G et al. Subcutaneous implantation of a new intravenous pump system for prostacyclin treatment in patients with pulmonary arterial hypertension. Heart Lung 2012 Aug 21. [Epub ahead of print]

Such pumps have been implanted in more than 90 patients in various European countries during the past 3 years. Experience shows that most of the patients selected for implantation have FC II-IV under combination therapy (2-3 specific PH-medications). The previous medication was either regarded as insufficient in respect to cardiopulmonary stabilization or the side effects of the therapy were intolerable. The latter applied particularly to patients with subcutaneous delivery of treprostinil in fairly large doses.

Given the previous application of the LENUS Pro® pump in the context of individualized healing attempts, the initiators of the planned study consider that it is necessary to ascertain the safety of this fully implantable pump system in a controlled prospective study.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

Patient aged ≥ 18 years Patient (or patient's legally authorized representative) is willing and able to provide written informed consent Patient is willing and able to comply with the protocol, including required follow-up visits Patient is diagnosed with Pulmonary Arterial Hypertension (World Health Organization (WHO) Category Group 1 (by the WHO Clinical classification system), including Idiopathic (IPAH), Heritable PAH (HPAH) (Familial PAH), and PAH associated with other diseases (APAH), Patient is receiving continuous infusion of treprostinil via subcutaneous or intravenous delivery using an external pump system Patient is in stable clinical condition und the previous specific PH medication has been retained unchanged during the past 3 weeks Patient's anticoagulation therapy can be managed to permit safe device implantation

Exclusion Criteria:

* Pregnancy, nursing Women of childbearing potential who are not on a reliable and safe form of contraception Patient is diagnosed with PH with an etiology different from that of the inclusion criteria, Patient is diagnosed with chronic kidney disease (estimated GFR <30) within ninety (90) days prior to Baseline visit; chronic kidney disease is defined as that lasting or expected to last more than three (3) months.

Hepatic insufficiency (Child C) Patient is a person whose body size is not sufficient to accept implantable pump bulk and weight as determined by the implanting surgeon Unacceptably high anesthetic risk as determined by the treating anesthesiologist Concomitant medication or underlying disease associated with an increased infection risk (e.g., intravenous drug abuse, diabetic gangrene) Patient is not in stable condition, especially a manifestation of decompensated right heart failure within three weeks prior to Baseline visit Patients with significantly increased bleeding risk due to comorbidities (e.g. hereditary F VIII deficiency, myeloproliferative neoplasm) Estimated life expectancy < 6 months due to comorbidities (e.g. terminal malignancy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from pulmonary centers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-04 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Measurement of numbers of predefined complications in longterm treatment with LenusPro medication pump | from implantation of pump (baseline) up to six month after implantation
  Rate and type of predefined intraoperative complications (by implantation) as assessed by the implanting physician:
Measurement of catheter (or pump) complications | from implantation of pump up to month six
  Rate and type of predefined catheter (or pump) complications

SECONDARY OUTCOMES:
Measurement of numbers of predefined refill complications | from implanation of pump (baseline) up to six month after implantation
  Refill complications, e.g. filling impossible because filling port cannot be found or fluoroscopy required to find filling port

OTHER OUTCOMES:
Measurement of quality of life (QoL) | from implantation of pump (baseline) up to six months after implantation
  Patient reported outcome (Questionaire EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Ewert, M.D., Principal Investigator — University Hospital of Greifswald
Locations (4):
- Krankenhaus der Elisabethinen Linz, Linz, Austria
- Germany (2):
  - University Hospital of Greifswald, Greifswald, Germany
  - Universitätsklinik Giessen, Giessen
- VU University Medical Center, Amsterdam, Netherlands